CLINICAL TRIAL: NCT03549884
Title: Delayed Cord Clamping in Infants Born by Cesarean Section: a Randomized Controlled Trial
Brief Title: Delayed Cord Clamping in Infants Born by Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4443/AO/18
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Umbilical Cord Management; Elective Cesarean Section
Keywords: Early cord Clamping; Delayed cord clamping; Full term infant; Elective cesarean section; Hematocrit; Postnatal adaptation
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The health care giver who will perform hematocrit measurement (primary outcome) and the statistician who will perform data analysis will be blind for treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed cord clamping (DCC) (Experimental): Cord clamping will be performed after 60 seconds of life
  Interventions: Procedure: Delayed cord clamping
- Early cord clamping (ECC) (Active Comparator): Cord clamping will be performed within 10 seconds of life
  Interventions: Procedure: Early cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — Cord clamping will be performed after 60 seconds of life in infants delivered by cesarean section
  Arms: Delayed cord clamping (DCC)
Procedure: Early cord clamping — Cord clamping will be performed within 10 seconds of life in infants delivered by cesarean section
  Arms: Early cord clamping (ECC)

SUMMARY:
Introduction: Placental transfusion supports an important blood transfer to the neonate, promoting a more stable and smooth transition from fetal to extra-uterine life. Cesarean section, especially elective one, reduces the placental transfusion, mainly because of uterine atony. Therefore, during an elective cesarean section umbilical cord management may play a relevant role on blood passage to the neonate and, as consequence, it may affect neonatal hematological values and cardiovascular parameters. The most effective way to manage umbilical cord in in elective cesarean section remains to be established.

Objective: The aim of the present study is to evaluate the effect of two different methods of umbilical cord management (Early Cord Clamping - ECC vs. Delayed Cord Clamping - DCC) on the hematocrit on the second day of life; in addition, we will assess the effect on perinatal and postnatal cardiovascular parameters.

Material and methods: This is a randomized clinical trial on the effect of different cord management newborns born by cesarean sections. After obtaining parental consent, all mothers > 38 weeks' gestation will be assigned to eithr ECC or DCC group in a 1:1 ratio according to a computer-generated randomized sequence. The primary outcome will be the hematocrit on day 2 of life. Secondary outcomes will be pre-ductal oxygen saturation (SaO2) and the heart rate (HR) during the first ten minutes after the birth, arterial blood pressures during the first 3 postnatal days and transcutaneous bilirubin (BT) at day 3 after birth.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section
* Gestational age > or = 39 weeks
* No labor
* Single pregnancy
* Parental consent; a written informed consent will be obtained by a member of the neonatal team involved in the study from a parent or guardian

Exclusion Criteria:

* Emergent or urgent cesarean sections
* Twin pregnancies
* Parental refusal to participate to the study
* Major congenital malformations (such as cardiopathies)
* Chromosomic abnormalities
* Fetal hydrops
* Severe maternal diseases (such as hypertension)
* Cord abnormalities (length < 20 cm, funicular prolapse, funicular knots)
* Intrauterine growth restriction (IUGR)

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Hematocrit | Day 2 of life

SECONDARY OUTCOMES:
Preductal transcutaneous saturation (TcSaO2) | During the first 10 minutes of life
Heart rate | During the first 10 minutes of life
  (bpm)
Arterial blood pressure | At day 1, 2, 3 of life
  (mmHg)
Total transcutaneous bilirubin | Day 3 of life
  (mg/dl)
Maternal blood losses | At delivery
  ml
Temperature at Normal nursery admission | At the time of normal nursery admission
  Celsius degrees
Time to the first breath | At birth
  seconds
Weight | Day 3 of life
  g

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Trevisanuto, MD, Principal Investigator — University of Padova, Italy
Locations (1):
- Azienda Ospedaliera di Padova, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2018
Access Criteria: Contacting PI by e-mail

REFERENCES:
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal Resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S204-41. doi: 10.1161/CIR.0000000000000276. No abstract available. PMID 26472855
- [Background] Katheria AC, Brown MK, Rich W, Arnell K. Providing a Placental Transfusion in Newborns Who Need Resuscitation. Front Pediatr. 2017 Jan 25;5:1. doi: 10.3389/fped.2017.00001. eCollection 2017. PMID 28180126
- [Background] Zhou YB, Li HT, Zhu LP, Liu JM. Impact of cesarean section on placental transfusion and iron-related hematological indices in term neonates: a systematic review and meta-analysis. Placenta. 2014 Jan;35(1):1-8. doi: 10.1016/j.placenta.2013.10.011. Epub 2013 Nov 20. PMID 24290868
- [Background] Erickson-Owens DA, Mercer JS, Oh W. Umbilical cord milking in term infants delivered by cesarean section: a randomized controlled trial. J Perinatol. 2012 Aug;32(8):580-4. doi: 10.1038/jp.2011.159. Epub 2011 Nov 17. PMID 22094494
- [Background] Fogarty M, Osborn DA, Askie L, Seidler AL, Hunter K, Lui K, Simes J, Tarnow-Mordi W. Delayed vs early umbilical cord clamping for preterm infants: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Jan;218(1):1-18. doi: 10.1016/j.ajog.2017.10.231. Epub 2017 Oct 30. PMID 29097178